CLINICAL TRIAL: NCT06572345
Title: A Multicentre Open-Label, Feasibility Study of the Use of a Short-Term Low-Energy Diet in Adolescents With Obesity and Type-2 Diabetes Mellitus
Brief Title: Low EnerGy DiEt iN Adolescents With Obesity and Type 2 Diabetes: The LEGEND Study
Acronym: LEGEND
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Collaborators: Diabetes UK (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22CS007; 21/0006341 (Other Grant/Funding Number: Diabetes UK); 317544 (Other: IRAS Number)
Record Dates: First submitted 2024-06-07; First posted 2024-08-27 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-08

CONDITIONS: Pediatric Obesity; Type 2 Diabetes
Keywords: Type 2 diabetes mellitus; Paediatric; Obesity; Low-energy diet; Adolescent; Remission
MeSH Terms: conditions — Pediatric Obesity; Diabetes Mellitus, Type 2; Obesity | interventions — Caloric Restriction

STUDY DESIGN:
Intervention Model Description: 73 participants in total:
  * Thirty-three participants to trial the LED intervention
  * Ten participants from the LED intervention and their parents/carers for the interviews.
  * Ten dyads undertaking interviews only (1 adolescent and 1 parent/carer) who declined the intervention.
  * Ten healthcare practitioners (interviews only).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Low Energy Diet (LED) (Experimental): 33 participants will undergo a 12 week low energy diet (LED), followed by a 12 week food reintroduction phase and 24 week weight maintenance phase. 10 participant across all sites from this intervention will be asked to complete a qualitative interview at 2 time points throughout the study, alongside their parent/carer, to understand their thoughts around the intervention, their experience taking part in the study and suggestions for improvement.
  Additionally, further interviews will be undertaken with participants and their relatives/carers who declined to take part in the LED portion of the study to understand the reasons why/barriers to them taking part in the intervention. Furthermore, 10 health care professionals (HCPs) from different sites involved in the study will be invited to take part in interviews to garner feedback and experience as well as their impression of the experience of the study for the participants and their families.
  Interventions: Dietary Supplement: Low-energy diet; Other: Qualitive interview - LED participants; Other: Qualitive interview - Participants declining LED; Other: Qualitive interview - Health Care Professionals (HCPs)

INTERVENTIONS:
Dietary Supplement: Low-energy diet — For the first 12 weeks during the LED, participants will have 4 meal replacement products each day. The following 12 weeks consists of a gradual reintroduction of food one meal at a time, in a structured stepwise progression, under the supervision of a dietitian. They will then undergo 28 weeks of weight maintenance to see if they are able to keep their weight stable.
Other: Qualitive interview - LED participants — Semi-structured interviews with 10 of the LED participants and their relative/carer.
Other: Qualitive interview - Participants declining LED — Semi-structured interviews with 10 participants who declined the LED, and their relative/carer.
Other: Qualitive interview - Health Care Professionals (HCPs) — Semi-structured interviews with 10 HCPs involved in delivery of the trial.

SUMMARY:
This is a multicentre, single-arm, feasibility study in adolescents with T2DM and obesity to investigate the recruitment and retention rates to a study using Low Energy Diets(LED). It will also provide estimates of weight loss needed to bring about remission to inform a larger randomised study. In addition a subgroup of participants and their parents/carers undertaking a period of LED will be interviewed to understand the participants experience of taking part. Two further groups will also be interviewed: participants and their parents/carers who have declined to take part in the LED to understand their motivations and barriers and healthcare practitioners who have participated in conducting the trial to understand their experience of the study.

DETAILED DESCRIPTION:
LED intervention

The three-stage intervention, will be delivered by the local study dietitian and doctor. Participants will typically undergo a 12-week intensive LED intervention followed by a 12-week Food Re-introduction (FR) phase and then a Weight Maintenance (WM) phase. The aim is for participants to lose 15kg (or 15% of starting body weight if<80kg at baseline) and achieve remission defined as an HbA1C <48 mmol/mol three months apart.

The LED phase consists of a total meal replacement (TMR) diet for 12 weeks which contains 800-1000cal/day (with LED diets typically containing 800-1200kcal/day), and has been previously shown to be safe in young people. Available products include shakes, soups and bars from providers such as Cambridge 1:1, Lighter Life and Optifast. TMR products will be supplied and distributed by the study team at no cost to the participant. The experience of other investigators suggests that having prepared shakes and bars reduces the anxiety associated with meal choices and preparation. If participants are not able to adhere to only four meal replacement products a day, a low-energy meal option for up to one meal a day (instead of a TMR product and using low-calorie recipes provided as part of the study) may be suggested and discussed by the research team.

Following the initial LED phase, participants will enter the FR phase, typically over the next 12 weeks. This consists of a gradual reintroduction of food one meal at a time, in a structured stepwise progression and under the supervision of a dietitian. A recipe book of 400-500 kcal recipes has been developed for this purpose.

If the target weight is achieved before 12 weeks, the FR phase may be brought forward.

If the HbA1C has fallen to below the pre-diabetes range (less than 42 mmol/mol) on point of care testing, but the target weight has not been achieved, FR phase may still be initiated at 12 weeks. If the target weight is not achieved by 12 weeks and the HbA1C remains 48 mmol/mol or above, the LED phase could be extended to a maximum of a total of 20 weeks duration, in discussion with the participant and the parents/carers, as appropriate.

If, during FR, the participant gains 2kg or more, there is flexibility to regress a step along the FR pathway, at the discretion of the local team and in discussion with the participant and their family, mirroring the successful pragmatic approach of the DiRECT study. For instance, a participant who has introduced their first meal and gains 2kg, may go back to full LED; someone who has gained weight after moving from two to three meals a day may go back to two meals. A participant who gains 2kg or more in the WM phase, may similarly go back one step to two meals a day. Locally, our experience using the LED showed the importance of a flexible approach, with some young people finding benefit from a short break (e.g. for a family celebration) or a preference to start during school holidays.

Current standard practice is to measure weight at each clinic with height and HbA1C checked once every 3 months. In addition to these routine measurements, data on participants' weight, height, HbA1C and adherence will be collected by the local diabetes team at each face-to-face visit and entered directly into the study data collection forms by either a study healthcare professional (HCP) or research nurse, as well as recorded in the participants medical record.

During the LED and FR phases, participants will have two-weekly clinical contact with face-to-face contact at least every four weeks which will include repeat anthropometry (including weight and blood pressure). Biochemistry will be repeated.

During the maintenance phase, contacts will aim to be every four weeks with no more than six weeks between contacts.

Participants' data will be collected by the local diabetes team or research nurses at each visit and recorded in the participants medical record. Data will be entered into the study approved electronic case-report form (CRF) system by the local diabetes or research teams.

Study questionnaires will be undertaken at baseline, during LED, during FR and in the follow-up period using an approved electronic CRF system by either the participant or research nurse. Physical activity assessment, MRI scans and dual x-ray anthropometry (DXA) scans will be undertaken at baseline, during the transition between phases and at the end of the study period. Physical activity level will be assessed by using activity trackers, six-minute walking test and a physical activity questionnaire. MRI scans will measure internal adipose deposits and DXA will measure fat and lean mass, bone mineral density and bone mineral content. Blood samples will be taken and analysed in local laboratories of units participating in the study. Results of tests undertaken locally will be entered on participants' CRF by the local research team.

Additional Interviews

Semi-structured interviews will be undertaken by a chartered clinical psychologist with a subset of the young people who took part in the LED intervention to understand the adolescents experience of taking part in the study midway through the study and at the end.

Semi-structured interviews will also be undertaken by a chartered clinical psychologist with 10 young people and/or their family who opted not to take part in the LED study to help understand barriers to participation and how these can be minimised.

Qualitative interviews will also be conducted with at least 10 healthcare professionals from different sites involved in the study to garner feedback and experience as well as the HCPs impression of the experience of the study for the participants and their families.

It is suggested that the proposed number of interview participants will be sufficient to meet the research aims. However, data saturation (whereby no new information is reported) will guide the recruitment process. In each case, purposefully constructed interview guides will be formulated to enhance the rigour of the data generated. All interviews will be conducted remotely with Hilton Health Consultancy via an approved platform. All interviews will be recorded and transcribed and analysed by Hilton Health Consultancy.

This feedback will be instrumental in informing and shaping any subsequent randomised control trial.

ELIGIBILITY:
Inclusion criteria

LED intervention

* Diagnosis of T2DM (defined as an HbA1C ≥48mmol/mol, in the absence of features of type 1 or monogenic/syndromic diabetes).
* Current HbA1C ≥48 (or ≥42 on antidiabetic medication) and ≤ 80 mmol/mol.
* Aged 12 to 17 years old.
* BMI ≥98th centile (+2 SD) for age and sex (UK90 growth reference data).
* Informed consent:

  * Received from the young person (age 16-17) OR
  * Received from young person's parent/carer, with patient assent (age 12-15).
* Willing to engage in and commit to low energy diet, FR and weight management phases including follow-up and attending study visits.

LED Intervention Interviews

The same interview inclusion criteria for LED intervention, with the following additional requirements:

Patients:

* Informed consent:

  * Received from the young person (age 16-17) OR
  * Received from young person's parent/carer, with patient assent (age 12-15).
* Willing to take part in a qualitative interview alongside a parent/carer.

Relative/Carer:

* A relative/carer for a young person meeting the above LED participant eligibility criteria.
* Informed consent from the relative/carer to participate in the interview.
* Willing to take part in a qualitative interview alongside the young person.

Non-LED Qualitative Interview only participants

* Diagnosis of T2DM (defined as an HbA1C ≥48mmol/mol, in the absence of features of type 1 or monogenic/syndromic diabetes).
* Current HbA1C ≥48 (or ≥42 on antidiabetic medication) and ≤80 mmol/mol.
* Aged 12 to 17 years old.
* BMI ≥98th centile (+2 SD) for age and sex (UK90 growth reference data).
* Informed consent:

  * Received from the young person (age 16-17) OR
  * Received from young person's parent/carer, with patient assent (age 12-15).
* Willing to take part in a qualitative interview alongside a parent/carer only.

HCPs

* Registered HCP.
* Experience of delivering this trial to the adolescents.
* Willing to take part in a qualitative interview about undertaking motivational interviewing training and conducting/delivering the LED intervention study.

Exclusion criteria

LED intervention

* HbA1C greater than 80mmol/mol.
* Presence of diabetes-related autoantibodies, as per local centre guidelines.
* Confirmed mono-genetic cause of obesity (e.g. SIM1 mutation) or diabetes-associated syndrome such as Prader-Willi syndrome, Bardet-Biedl or Wolfram's syndrome.
* Secondary diabetes (post bone marrow transplant/chemotherapy).
* Significant psychiatric co-morbidity.
* Breastfeeding, pregnant or planning to conceive during the LED and FR phases (female participants will be advised on need for effective contraceptive methods during the 12-month study period, section 5.1.1.10).
* Any other condition which, in the opinion of the study investigator, would make it inappropriate to undertake a period of LED. (All reasons for not approaching patients will be recorded and analysed anonymously. Cases can be discussed with the core study group if there is doubt).
* Participation in another interventional trial within 6 months.
* Informed consent and/or assent not received.
* Pre-existing retinopathy.
* Dietary avoidance (including, but not limited to, due to allergies, intolerances, religious reasons and lifestyle choices) to any ingredients in the meal replacement products, including lactose.
* Previous scoliosis repair.

Non-LED Qualitative Interview only participants

* HbA1C greater than 80mmol/mol.
* Presence of diabetes-related autoantibodies, as per local centre guidelines.
* Confirmed mono-genetic cause of obesity (e.g. SIM1 mutation) or diabetes-associated syndrome such as Prader-Willi syndrome, Bardet-Biedl or Wolfram's syndrome.
* Secondary diabetes (post bone marrow transplant/chemotherapy).
* Significant psychiatric co-morbidity.
* Breastfeeding, pregnant or planning to conceive during the LED and FR phases (female participants will be advised on need for effective contraceptive methods during the 12-month study period, section 5.1.1.10).
* Any other condition which, in the opinion of the study investigator, would either make it inappropriate to undertake a period of LED. (All reasons for not approaching patients will be recorded and analysed anonymously. Cases can be discussed with the core study group if there is doubt).
* Participation in another interventional trial within 6 months.
* Informed consent and/or assent not received.
* Pre-existing retinopathy.
* Dietary avoidance (including, but not limited to, due to allergies, intolerances, religious reasons and lifestyle choices) to any ingredients in the meal replacement products, including lactose.
* Previous scoliosis repair.

HCPs

• None.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 73 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of potential participants that can be recruited to an LED intervention | 12 months
  Number of eligible participants identified compared to those consented, passed screening and started on LED intervention.
Retention rate measured by by data availability for participant height. | 12 months
  Height obtained for the participant at:
  1. End of LED phase (12 weeks)
  2. End of FR phase (24 weeks)
  3. End of maintenance phase (12 months)
Retention rate measured by by data availability for participant weight. | 12 months
  Weight obtained for the participant at:
  1. End of LED phase (12 weeks)
  2. End of FR phase (24 weeks)
  3. End of maintenance phase (12 months)
Retention rate measured by by data availability for participant HbA1C. | 12 months
  HbA1C obtained for the participant at:
  1. End of LED phase (12 weeks)
  2. End of FR phase (24 weeks)
  3. End of maintenance phase (12 months)

SECONDARY OUTCOMES:
Proportion of participants that adhere to the LED | 12 weeks
  Defined by at least 5% weight loss at end of LED phase compared to baseline.
Degree of weight loss achieved in those who adhere to the LED and if this is maintained at 12-months. | 12 months
  Weight as measured at end of LED phase (12 weeks), compared against weight as measured at baseline.
  Weight as measured at end of FR phase (24 weeks), compared against weight as measured at baseline.
  Weight as measured at end of maintenance (12 months) compared against weight at baseline.
  Weight as measured at end of FR compared against weight at the end of LED phase.
  Weight as measured at end of maintenance (12 months) compared against weight at the end of LED phase.
Do those who adhere to the LED achieve remission? To determine the standard deviation of the proportion of participants that achieve remission (to estimate the sample size for a definitive randomised trial). | 12 months
  Percentage weight loss in those who achieve remission of T2DM defined as an HbA1C <48 mmol/mol on two occasions at least 3 months apart, in the absence of anti-diabetes medication. This will help to determine the standard deviation of the proportion of participants that achieve remission, to enable an estimation of sample size for a future, definitive, randomised control trial.
Do those who adhere to the LED achieve remission? To determine the standard deviation of the proportion of participants that achieve remission (to estimate the sample size for a definitive randomised trial). | 12 months
  Absolute weight loss in those who achieve remission of T2DM defined as an HbA1C <48 mmol/mol on two occasions at least 3 months apart, in the absence of anti-diabetes medication. This will help to determine the standard deviation of the proportion of participants that achieve remission, to enable an estimation of sample size for a future, definitive, randomised control trial.
Adverse effects | 12 months
  Collection of adverse events at every study visit.
Is the study, including the intervention, investigations and assessments, deliverable consistently across different sites using the standardised study resources. | 12 months
  Qualitative interviews with patients and carers (patient and carers interviewed together) who participate in the LED, and those who do not.
Is the study, including the intervention, investigations and assessments, deliverable consistently across different sites using the standardised study resources. | 12 months
  Qualitative interviews with healthcare professionals who are involved in delivering the study.
Which biomarkers and pathways are upregulated and which are downregulated in young people with T2DM and what is the response to an LED intervention. | 12 months
  Understanding the pattern of and metabolic changes in:
  • water soluble metabolites before (at baseline) and after following a LED (at end of LED - 12 weeks, end of FR -24 weeks and end of WM - 12 months).
Which biomarkers and pathways are upregulated and which are downregulated in young people with T2DM and what is the response to an LED intervention. | 12 months
  Understanding the pattern of and metabolic changes in:
  • lipid metabolites before (at baseline) and after following a LED (at end of LED - 12 weeks, end of FR -24 weeks and end of WM - 12 months).
What are the positive and potential negative effects of a period of LED on the biological wellbeing of adolescents. | 12 months
  Changes in clinical markers, such as blood pressure, including both systolic and diastolic measurements (mmHg).
What are the positive and potential negative effects of a period of LED on the biological wellbeing of adolescents. | 12 months
  HbA1C
What are the positive and potential negative effects of a period of LED on the biological wellbeing of adolescents. | 12 months
  Full Blood Count
What are the positive and potential negative effects of a period of LED on the biological wellbeing of adolescents. | 12 months
  Ferritin
What are the positive and potential negative effects of a period of LED on the biological wellbeing of adolescents. | 12 months
  White Blood Cell Count
What are the positive and potential negative effects of a period of LED on the biological wellbeing of adolescents. | 12 months
  Platelet count
What are the positive and potential negative effects of a period of LED on the biological wellbeing of adolescents. | 12 months
  Urea and electrolytes
What are the positive and potential negative effects of a period of LED on the biological wellbeing of adolescents. | 12 months
  alanine transaminase (ALT)
What are the positive and potential negative effects of a period of LED on the biological wellbeing of adolescents. | 12 months
  Aspartate Transferase (AST)
What are the positive and potential negative effects of a period of LED on the biological wellbeing of adolescents. | 12 months
  Gamma Glutamyl Transferase (GGT)
What are the positive and potential negative effects of a period of LED on the biological wellbeing of adolescents. | 12 months
  Albumin
What are the positive and potential negative effects of a period of LED on the biological wellbeing of adolescents. | 12 months
  Lipid Profile - Cholesterol, triglycerides, low density lipoprotein, high density lipoprotein (all mg/DL)
What are the positive and potential negative effects of a period of LED on the biological wellbeing of adolescents. | 12 months
  Bone profile - Parathyroid hormone (PTH)
What are the positive and potential negative effects of a period of LED on the biological wellbeing of adolescents. | 12 months
  Bone profile - Calcium and Phosphate (mmol)
What are the positive and potential negative effects of a period of LED on the biological wellbeing of adolescents. | 12 months
  Bone profile - Alkaline Phosphatase (ALP) (U/L)
What are the positive and potential negative effects of a period of LED on the biological wellbeing of adolescents. | 12 months
  Bone profile - Vitamins A and E (ummol/L)
What are the positive and potential negative effects of a period of LED on the biological wellbeing of adolescents. | 12 months
  Bone profile - Vitamin D (nmol/L)
What are the positive and potential negative effects of a period of LED on the biological wellbeing of adolescents. | 12 months
  Thyroid function tests - T3 and T4 (pmol/L)
What are the positive and potential negative effects of a period of LED on the biological wellbeing of adolescents. | 12 months
  Thyroid function tests - Thyroid Stimulating Hormone (TSH) (mU/L)
What are the positive and potential negative effects of a period of LED on the biological wellbeing of adolescents. | 12 months
  luteinizing hormone (LH), follicle stimulating hormone (FSH) (u/L)
What are the positive and potential negative effects of a period of LED on the biological wellbeing of adolescents. | 12 months
  Testosterone, sex hormone binding globulin (nmol/L)
What are the positive and potential negative effects of a period of LED on the biological wellbeing of adolescents. | 12 months
  Oestradiol (pmol/L)
What are the positive and potential negative effects of a period of LED on the biological wellbeing of adolescents. | 12 months
  Changes in imaging markers such as liver fat on MRI
What are the positive and potential negative effects of a period of LED on the biological wellbeing of adolescents. | 12 months
  Changes in metabolic disease based on DXA scan
What are the positive and potential negative effects of a period of LED on the biological wellbeing of adolescents. | 12 months
  Changes in bone mineral density based on DXA scan
What are the positive and potential negative effects of a period of LED on the biological wellbeing of adolescents. | 12 months
  Changes in body composition based on DXA scan
What are the positive and potential negative effects of a period of LED on the psychological wellbeing of adolescents. | 12 months
  Change in eating disorder score or development of eating disorders and binge eating, assessed via the Eating Disorder Examination Questionnaire EDE-Q/EDE-A.
What are the positive and potential negative effects of a period of LED on the psychological wellbeing of adolescents. | 12 months
  Change in psychological outcomes via the Generalised Anxiety Disorder Assessment (GAD-7).
What are the positive and potential negative effects of a period of LED on the psychological wellbeing of adolescents. | 12 months
  Change in psychological outcomes via the Revised Children's Anxiety and Depression Scale (RCAS).
What are the positive and potential negative effects of a period of LED on the social wellbeing of adolescents. | 12 months
  Change in health-related quality of life via Child Health Utility instrument (CHU9D).
What are the positive and potential negative effects of a period of LED on the social wellbeing of adolescents. | 12 months
  Change in health-related quality of life via the paediatric quality of life inventory - PedsQL 3.2.
What are the positive and potential negative effects of a period of LED on the social wellbeing of adolescents. | 12 months
  Change in health-related quality of life via EQ-5D-Y, a standardised measure adapted for use with young people.
What are the positive and potential negative effects of a period of LED on the behavioural wellbeing of adolescents. | 12 months
  Change in activity via activity monitors.
What are the positive and potential negative effects of a period of LED on the behavioural wellbeing of adolescents. | 12 months
  Change in activity through self-report via Physical Activity Questionnaire (PAQ-A/PAQ-C).
What are the positive and potential negative effects of a period of LED on the behavioural wellbeing of adolescents. | 12 months
  Acceptability of the intervention from semi-structured interviews conducted with participants and their family/carer, simultaneously.

CONTACTS AND LOCATIONS:
Locations (1):
- Nottingham University Hospital NHS Trust, Nottingham, United Kingdom